CLINICAL TRIAL: NCT00536315
Title: Tracheal Mechanics During Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Loring, Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2001P001418
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2010-02

CONDITIONS: Tracheomalacia; Tracheobronchomalacia
Keywords: COPD
MeSH Terms: conditions — Tracheomalacia; Tracheobronchomalacia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- COPD: Patients with cough and/or shortness of breath who may have windpipe collapse.
- Healthy adults: Subjects without symptoms for comparison.
- Tracheomalacia: Patients with cough and/or shortness of breath who may have windpipe collapse.

SUMMARY:
The main purpose of this study is use a new type of measurement to help decide what kind of therapy would help people with a collapsing windpipe or tracheomalacia.

DETAILED DESCRIPTION:
This study is to obtain new information about the pressures required to collapse the trachea in patients with and without obstructive pulmonary disease and to describe the relationship between pressures and airflow obstruction. This information will provide normative data not currently available and would establish whether tracheal collapse is due to tracheomalacia. The data may lead to better ways of predicting if a patient would benefit from procedures to prevent tracheal collapse.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of tracheal collapse undergoing bronchoscopy
* Healthy control subject undergoing bronchoscopy for another purpose.

Exclusion Criteria:

* Esophageal pathology
* Tracheostomy
* inability to follow commands

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy control subjects recruited from subjects volunteering for CT or bronchoscopic studies and patients referred for evaluation of possible tracheomalacia.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 1999-03-01 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Loring, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Loring SH, O'donnell CR, Feller-Kopman DJ, Ernst A. Central airway mechanics and flow limitation in acquired tracheobronchomalacia. Chest. 2007 Apr;131(4):1118-24. doi: 10.1378/chest.06-2556. PMID 17426218